CLINICAL TRIAL: NCT01916499
Title: MRI Study After Arterial Switch Operation in Patients With Transposition of the Great Arteries
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kathrine Rydén Suther, MD, Oslo University Hospital
Other Study IDs: 2011/1422
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Transposition of Great Vessels; Surgery
Keywords: Child, adolescent; Coronary artery disease; Magnetic resonance imaging
MeSH Terms: conditions — Transposition of Great Vessels; Coronary Artery Disease | interventions — Ventricular Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Switch "trap-door" re-implantation of the coronaries: Re-implantation of the coronary arteries into the neo-aortic sinuses through a "trap-door" as far distally as possible on the neo-aorta
  Interventions: Other: 3 tesla magnetic resonance imaging findings; coronary artery status; Other: 3 tesla magnetic resonance imaging findings; ventricular function and morphology
- Switch non-"trap-door" re-implantation of the coronaries: Re-implantation of the coronary arteries into the neo-aortic sinuses through small incisions or excision in the sinuses
  Interventions: Other: 3 tesla magnetic resonance imaging findings; coronary artery status; Other: 3 tesla magnetic resonance imaging findings; ventricular function and morphology

INTERVENTIONS:
Other: 3 tesla magnetic resonance imaging findings; coronary artery status
Other: 3 tesla magnetic resonance imaging findings; ventricular function and morphology

SUMMARY:
This study involves adolescents operated with arterial switch procedure for transposition of the great arteries during the neonatal period. The purpose is to evaluate the coronary arteries and direct and indirect findings of coronary artery disease/complications with 3 tesla magnetic resonance imaging.

DETAILED DESCRIPTION:
This study involves adolescents operated with arterial switch procedure for transposition of the great arteries during the neonatal period. The patients were operated with two different methods of re-implantation of the coronary arteries ("trap-door"/non-"trap-door", see description below).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of transposition of the great arteries with or without ventricular septum defect
* Surgically corrected during neonatal period with arterial switch procedure

Partial or total Exclusion Criteria:

* Heart arrhythmias
* Known allergic reaction to gadolinium based contrast media
* Reduced renal function (below 60 ml/min/1,73m2)

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 10-15 years old surgically corrected in the neonatal period with arterial switch procedure for transposition of the great arteries at Rikshospitalet, OUS, Norway.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Direct visualization and status of the coronary arteries, global volume measurements, global and regional strain (myocardial contractility), extravascular, extracellular tissue volume fraction and late enhancement (myocardial fibrosis). | 10-15 years after surgery

SECONDARY OUTCOMES:
Comparison of image quality of direct visualization of the coronary arteries with and without contrast enhanced techniques. | 10-15 years after surgery
Comparison of coronary artery findings corresponding to indirect functional and morphological findings in MRI and echocardiography in the left and right ventricle. | 10-15 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte De Lange, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided